CLINICAL TRIAL: NCT03279120
Title: Phase I, 90-Day Safety, Pharmacokinetic, And Pharmacodynamic Study Of Intravaginal Rings Releasing Tenofovir And Levonorgestrel
Brief Title: Safety, PK, and PD Study of IVRs Releasing TFV and LNG
Acronym: TFV/LNG IVR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Agility Clinical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A15-138
Record Dates: First submitted 2017-08-23; First posted 2017-09-12 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Anti-Infective Agents; Anti-Retroviral Agents; Contraceptive Usage
Keywords: HIV; LNG; TFV; IVR; Contraception; Prevention
MeSH Terms: conditions — Contraception Behavior | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TFV/LNG IVR (8-10mg/20μg) (Continuous) (Experimental): TFV/LNG IVR is an intravaginal ring 55.0 mm in diameter, consisting of two segments of polyurethane tubing with an outer cross-sectional diameter of 5.5 mm: a longer segment (135 mm) containing white to off-white TFV paste and a shorter one (34 mm) with a translucent LNG core. Used for 90 days (continuous).
  Interventions: Drug: TFV/LNG IVR
- TFV/LNG IVR (8-10mg/20μg) (Interrupted) (Experimental): TFV/LNG IVR is an intravaginal ring 55.0 mm in diameter, consisting of two segments of polyurethane tubing with an outer cross-sectional diameter of 5.5 mm: a longer segment (135 mm) containing white to off-white TFV paste and a shorter one (34 mm) with a translucent LNG core. Used for 90 days (3x28 days interrupted).
  Interventions: Drug: TFV/LNG IVR
- Placebo (Continuous) (Placebo Comparator): Intravaginal ring 55.0 mm in diameter, consisting of two segments of polyurethane tubing with an outer diameter of 5.5 mm containing no active experimental ingredients. Used for one month. Used for 90 days (continuous).
  Interventions: Drug: Placebo
- Placebo (Interrupted) (Placebo Comparator): Intravaginal ring 55.0 mm in diameter, consisting of two segments of polyurethane tubing with an outer diameter of 5.5 mm containing no active experimental ingredients. Used for one month. Used for 90 days (3x28 days interrupted).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TFV/LNG IVR — Used for 90 days (Continuous or Interrupted)
  Other Names: Tenofovir/Levonorgestrel Intravaginal Ring
  Arms: TFV/LNG IVR (8-10mg/20μg) (Continuous); TFV/LNG IVR (8-10mg/20μg) (Interrupted)
Drug: Placebo — Used for 90 days (Continuous or Interrupted)
  Arms: Placebo (Continuous); Placebo (Interrupted)

SUMMARY:
This multi-center Phase I study is designed to characterize the safety, PK, and PD of TFV/LNG IVR to assess systemic and genital tract bioavailability in healthy women. The IVRs to be used in the study are TFV/LNG IVR (8-10mg per day/20μg per day) or placebo IVR. Samples will be obtained before, during and after 90 days of continuous or interrupted IVR use.

DETAILED DESCRIPTION:
The purpose of this multi-center Phase I protocol, titled Phase I, 90-Day Safety, Pharmacokinetic, and Pharmacodynamic Study of Intravaginal Rings Releasing Tenofovir and Levonorgestrel is to assess the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of the Tenofovir/Levonorgestrel Intravaginal Ring (TFV/LNG IVR).

The study will enroll healthy, non-pregnant, ovulatory, HIV-uninfected women aged 18 to 50 with a body mass index (BMI) less than 30 kg/m2, regular menstrual cycles (approximately 26-35 days) by participant report, and willing to use non-spermicidal condoms for sex and follow other study restrictions. Women will be protected from pregnancy by abstinence from vaginal intercourse or agreeing to consistently use condoms.

The enrollment goal is for approximately 60 participants to complete the study. A subset of approximately 20 women will be selected for an in-depth interview to take place during the first month of IVR use and again after 90 days of use.

Women will be randomized to one of four arms: TFV/LNG IVR (8-10mg per day/20μg per day) for 90 days (Continuous), TFV/LNG IVR (8-10mg per day/20μg per day) for 3x28 days (Interrupted), placebo IVR for 90 days (Continuous), or placebo IVR for 3x28 days (Interrupted) and will undergo blood, cervicovaginal and rectal fluid sample collections, and cervicovaginal tissue collections for PK and PD assessments before, during and after 90 days of continuous or interrupted IVR use.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-50 years, inclusive
* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes) and with an intact gastrointestinal tract, uterus, and cervix.
* Currently having regular menstrual cycles (approximately 26-35 days) by participant report
* History of Pap smears and follow-up consistent with standard clinical practice as outlined in the Study Manual or willing to undergo a Pap smear at Visit 1
* Protected from pregnancy by one of the following:
* Sterilization of either partner
* Abstinence from vaginal intercourse
* Consistent use of non-spermicidal condoms
* Willing to abstain from use of vaginal products (other than the study product and condoms) including tampons (except for menses), spermicides, lubricants, and douches for the whole study
* Willing to abstain from any vaginal and anal intercourse/activity starting 48 hours before cervical mucus collection, as possible, and 48 hours before Visits 4 and 29, and for 5 days after tissue collection
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection
* Negative urine pregnancy test
* P4 ≥3 ng/ml
* Willing to give voluntary consent and sign an informed consent form
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* BMI ≥ 30 kg/m2
* History of hysterectomy
* Currently pregnant or within two calendar months from the last pregnancy outcome.

Note: If recently pregnant, must have had at least two spontaneous menses since pregnancy outcome

* Use of any hormonal contraceptive method in the last 3 months (oral, transdermal, transvaginal, implant, or hormonal intrauterine contraceptive device)
* Injection of Depo-Provera in the last 10 months
* Use of copper IUD
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the study products, topical anesthetic, or to both silver nitrate and Monsel's solution
* Contraindication to LNG
* In the last three months, diagnosed with or treated for any STI or pelvic inflammatory disease. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility.
* Nugent score greater than or equal to 7 or symptomatic bacterial vaginosis (BV) as defined by Amsel's criteria
* Positive test for Trichomonas vaginalis (TV), Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), HIV-1, or Hepatitis B surface antigen (HBsAg)
* Known bleeding disorder, including deep vein thrombosis (DVT) and pulmonary embolism (PE), or those that could lead to prolonged or continuous bleeding with biopsy
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
* Known current drug or alcohol abuse which could impact study compliance
* Grade 2 or higher laboratory abnormality, per the 2014 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, or antivirals or antiretrovirals (e.g. acyclovir, valacyclovir, Viread®, Atripla®, Emtriva®, or Complera®), or CYP3A4 inducers or inhibitors as detailed in the Study Manual (e.g., St. John's Wort or erythromycin).

Note: Participants should avoid non-steroidal anti-inflammatory drugs (NSAIDs) except for treatment of dysmenorrhea during menses. Participants may use acetaminophen on an as-needed but not daily basis during the study.

* Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina, or cervix within the last 14 days
* Abnormal finding on laboratory or physical examination or a social or medical condition in the volunteer which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Percentage of women with Treatment-emergent adverse events | Day 90
  Treatment-emergent adverse events (TEAEs)
Changes in systemic laboratory values | Change from Baseline at Day 90
  Systemic laboratory values
Changes in cervicovaginal mucosa by visual inspection | Change from Baseline at Day 90
  Mucosal safety
Changes in soluble markers | Change from Baseline at Day 90
  Soluble markers in cervicovaginal fluid
Changes in inflammatory markers in cervicovaginal tissue | Change from Baseline at Day 90
  Inflammatory markers in cervicovaginal tissue
Changes in endogenous vaginal bacteria | Change from Baseline at Day 90
  Endogenous vaginal bacteria in cervicovaginal fluid
Microbial growth | Day 90
  Microbial growth on returned IVRs

SECONDARY OUTCOMES:
Maximum Plasma Concentrations [Cmax] | Baseline, 8 hours post-IVR insertion, Day 2 or 3 or 4 (randomized time point), 10, 21, 28, 32, 42, 53, 59, 63, 73, 84, 90; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Maximum Plasma Concentrations [Cmax] of TFV and LNG
Maximum CV Fluid Concentrations | 2 and 8 hours post-IVR insertion, Day 2 or 3 or 4 (randomized time point), 10, 21, 32, 42, 53, 63, 73, 84; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Maximum CV Fluid Concentrations of TFV
Maximum Rectal Fluid Concentrations | Day 2 or 3 or 4 (randomized time point), 21, 53, 84; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Maximum Rectal Fluid Concentrations of TFV
Maximum CV Tissue Concentrations | Changes from baseline at day 90; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Maximum CV Tissue Concentrations of TFV
Maximum CV Tissue Metabolite Concentrations | Changes from baseline at day 90; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Maximum CV Tissue Concentrations of TFV-DP
Maximum Serum Concentrations of LNG | Baseline, 1, 2, 4, and 8 hours post-IVR insertion, Day 2 or 3 or 4 (randomized time point), 10, 21, 28, 32, 42, 53, 59, 63, 73, 84, 90; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Maximum Serum Concentrations of LNG
Residual Drug Concentrations | Day 90
  Residual drug (TFV and LNG) in returned IVRs
Surrogates of contraceptive efficacy of Mucus | Day 30
  Surrogates of contraceptive efficacy: Cervical mucus assessment (Cervical mucus quality [score of >10])
Surrogates of contraceptive efficacy of Sperm | Day 30
  Surrogates of contraceptive efficacy: Cervical mucus assessment (Sperm migration on the Simplified Slide test)
Ovulation | Changes from baseline at day 90
  Ovulation by serum progesterone (P4)
Follicular Development | Changes from baseline at day 90
  Effect on follicular development by serum estradiol concentration
Antiviral activity in CV Fluid--HIV | Changes from baseline at day 90
  Anti-HIV-1 activity in CV fluid
Antiviral activity in CV Fluid--HSV-2 | Changes from baseline at day 90
  Anti-HSV-2 activity in CV fluid
Changes in Antiviral Activity | Changes from baseline at day 90
  Comparison of HIV-1 ex vivo infection in CV tissue (EVMS only) at baseline and after 90 days of IVR use
Bleeding Patterns | Baseline through Day 90 of IVR use
  Participant self-report of bleeding
Forgiveness--LNG | Day 32 and 63; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Decay of LNG during 3-day periods of non-use in interrupted regimen, and after 90 days of IVR use
Forgiveness--TFV | Day 32 and 63; and 48 or 72 hours or 5 days after IVR removal (randomized time point)
  Decay of TFV during 3-day periods of non-use in interrupted regimen, and after 90 days of IVR use
Acceptability--Qualitative | Baseline, Day 28 and 90
  Responses to key questions on acceptability and psychosocial questionnaire(s) (all participants), and feedback during in-depth interviews (subset of participants)
Acceptability--IDI | During first month of IVR use and Day 90
  Responses to key questions on acceptability and psychosocial questionnaire(s) (all participants), and feedback during in-depth interviews (subset of participants)
Adherence | Baseline, Day 28 and 90
  Percentage of participants with Discontinuations/Expulsions/Removals by self-report

OTHER OUTCOMES:
Antiviral activity in Rectal Fluid--HIV | Changes from baseline at day 90
  Anti-HIV-1 activity in rectal fluid
Antiviral activity in Rectal Fluid--HSV-2 | Changes from baseline at day 90
  Anti-HSV-2 activity in rectal fluid
Changes in Antiviral Activity--HSV-2 | Changes from baseline at day 90
  Comparison of HSV-2 ex vivo infection in CV tissue (EVMS-only) at baseline and after 90 days of IVR use, as possible
Qualitative TFV measurement | Day 90
  Qualitative measure of TFV in a vaginal swab
Adherence Marker in returned vaginal ring-analytic | Day 90
  Analytical measures of drug or placebo products
Adherence marker in returned ring--bioassay | Day 90
  Characterization of returned IVRs (active and placebo) via objective IVR biomarkers (e.g., residual glycerin content and bioassay) and residual drug (TFV and LNG), as feasible
Adherence marker in returned ring--correlation | Day 90
  Correlation of IVR removal scale factors and objective biomarkers of IVR use
Adherence marker in returned ring--correlation | Day 90
  Correlation of baseline user characteristics and objective biomarkers of IVR use

CONTACTS AND LOCATIONS:
Overall Officials: study director, Study Director — CONRAD
Locations (2):
- Eastern Virginia Medical School, Norfolk, Virginia, United States
- Profamilia, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurman AR, Brache V, Cochon L, Ouattara LA, Chandra N, Jacot T, Yousefieh N, Clark MR, Peet M, Hanif H, Schwartz JL, Ju S, Marzinke MA, Erikson DW, Parikh U, Herold BC, Fichorova RN, Tolley E, Doncel GF. Randomized, placebo controlled phase I trial of the safety, pharmacokinetics, pharmacodynamics and acceptability of a 90 day tenofovir plus levonorgestrel vaginal ring used continuously or cyclically in women: The CONRAD 138 study. PLoS One. 2022 Oct 10;17(10):e0275794. doi: 10.1371/journal.pone.0275794. eCollection 2022. PMID 36215267
- [Derived] Tolley EE, Zissette S, Taylor J, Hanif H, Ju S, Schwarz J, Thurman A, Tyner D, Brache V, Doncel GF. Acceptability of a Long-Acting, Multipurpose Vaginal Ring: Findings from a Phase I Trial in the U.S. and Dominican Republic. J Womens Health (Larchmt). 2022 Sep;31(9):1343-1352. doi: 10.1089/jwh.2021.0394. Epub 2022 Apr 1. PMID 35363574
- [Derived] Thurman AR, Ravel J, Gajer P, Marzinke MA, Ouattara LA, Jacot T, Peet MM, Clark MR, Doncel GF. Vaginal Microbiota and Mucosal Pharmacokinetics of Tenofovir in Healthy Women Using a 90-Day Tenofovir/Levonorgestrel Vaginal Ring. Front Cell Infect Microbiol. 2022 Mar 8;12:799501. doi: 10.3389/fcimb.2022.799501. eCollection 2022. PMID 35350436